CLINICAL TRIAL: NCT00689156
Title: Randomized Trial of Epirubicin and Cyclophosphamide Followed by Docetaxel Against Docetaxel and Cyclophosphamide in Patients With TOP2A Normal Early Breast Cancer
Brief Title: Epirubicin or Not in Patients With TOP2A (Topoisomerase (DNA) II Alpha (170kD)) Normal Early Breast Cancer
Acronym: READ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: Fonden Til Fremme af Klinisk- Eksperimentel Cancerforskning (Other); Sanofi (Industry); Dako (Industry)
Responsible Party: Principal Investigator, Bent Ejlertsen, Professor, MD, PhD, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG 07-READ
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-01

CONDITIONS: Breast Neoplasms
Keywords: Epirubicin; docetaxel; Adjuvant chemotherapy; DNA Topoisomerases, Type II
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen 1 (Active Comparator): Epirubicin 90 mg/m2 plus cyclophosphamide 600 mg/m2 intravenously day 1 every 3 weeks times three followed by docetaxel 100 mg/m2 intravenously day 1 every 3 weeks times three
  Interventions: Drug: Epirubicin, cyclophosphamide and docetaxel
- Regimen 2 (Experimental): Docetaxel 75 mg/m2 plus cyclophosphamide 600 mg/m2 intravenously day 1 every 3 weeks times six
  Interventions: Drug: docetaxel, cyclophosphamide

INTERVENTIONS:
Drug: Epirubicin, cyclophosphamide and docetaxel — Epirubicin 90 mg/m2 iv day 1 every 3 weeks plus Cyclophosphamide 600 mg/m2 iv day 1 every 3 weeks times 3 followed by Docetaxel 100 mg/m2 iv day 1 every 3 weeks times 3
  Other Names: Ellence; Taxotere
  Arms: Regimen 1
Drug: docetaxel, cyclophosphamide — Docetaxel 75 mg/m2 plus cyclophosphamide 600 mg/m2 intravenously day 1 every 3 weeks times six
  Other Names: Taxotere
  Arms: Regimen 2

SUMMARY:
The Danish Breast Cancer Cooperative Group (DBCG) wishes to clarify if recurrence-free and overall life expectancy is longer after docetaxel and cyclophosphamide compared to epirubicin and cyclophosphamide followed by docetaxel in patients with TOP2A normal and operable breast cancer.

DETAILED DESCRIPTION:
In DBCG trial 89D we in more than 1,200 patients showed that substitution in CMF chemotherapy of methotrexate with epirubicin improves survival for patients with primary and operable breast cancer. In a retrospective evaluation we have also shown that approximately 20% of all patients in 89D have tumors with numerical changes of the TOP2A gene, and that only patients with abnormal TOP2A benefit from epirubicin. In the current trial the DBCG wishes to clarify if recurrence-free and overall life expectancy is longer after docetaxel and cyclophosphamide compared to epirubicin and cyclophosphamide followed by docetaxel in patients with TOP2A normal and operable breast cancer.

ELIGIBILITY:
Trial Population:

1. Younger than 35, but at least 18 years of age
2. Hormone receptor-negative tumor (ER- and PgR-negative) and 35 to 75 years of age.
3. Hormone receptor-positive tumor, 35 to 59 years of age and presenting at least one of the following characteristics: spread to lymph nodes, tumor > 2 cm, degree of malignancy II-III or HER2-positive.

Inclusion Criteria:

1. Signed informed consent
2. Histologically confirmed invasive breast carcinoma which has been micro-radical removed by breast preserving surgery or mastectomy according to DBCG's guideline
3. TOP2A normal tumor (score of 0.8 - 2.0)

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Earlier medical cancer treatment, including docetaxel, epirubicin or cyclophosphamide.
3. Distant metastases or bilateral breast cancer (excluded after checking by means of chest radiography, bilateral mammography and normal blood samples as a minimum).
4. Other active, malign disease in the latest 5 years, except for adequately treated and cured carcinoma in situ cervices uteri or non-melanoma skin cancer.
5. Comorbidity score > 3 (patients with a score of 1-2 start at dose level -1).
6. Treatment with a non-approved product or test product in the latest 30 days.
7. Known severe hypersensitivity to docetaxel, epirubicin or cyclophosphamide or auxiliary agents in these products.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2015 (Actual)
Dates: Start 2008-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
IDFS; invasive disease-free survival | Within 10-yeras

SECONDARY OUTCOMES:
Overall survival | Life-long observation
DDFS; distant disease-free survival | Within 10-years
Serious adverse events | Within 10-years

CONTACTS AND LOCATIONS:
Overall Officials: Bent Ejlertsen, M.D., Principal Investigator — Rigshospitalet, Denmark; Henning T. Mouridsen, M.D., Study Director — Rigshospitalet, Denmark
Locations (13):
- Denmark (13):
  - Dept. of Oncology; Aalborg Sygehus, Aalborg
  - Dept. of Oncology; Århus Sygehus, Aarhus
  - Dept. of Oncology; Rigshospitalet, Copenhagen
  - Dept. of Oncology; Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Dept. of Oncology; Herlev Hospital, Herlev
  - Dept. of Oncology; Regionshospitalet Herning, Herning
  - Dept. of Oncology; Nordsjællands Hospital Hillerød, Hillerød
  - Dept. of Oncology; Sygehus Syd Næstved, Næstved
  - Dept. of Oncology; Odense University Hospital, Odense
  - Dept. of Oncology; Sygehus Øst Roskilde, Roskilde
  - Dept. of internal medicine; Bornholms Hospital, Rønne
  - Dept. of Oncology; Vejle Sygehus, Vejle
  - Dept. of Oncology; Regionshospitalet Viborg, Viborg

REFERENCES:
- [Background] Moller S, Jensen MB, Ejlertsen B, Bjerre KD, Larsen M, Hansen HB, Christiansen P, Mouridsen HT; Danish Breast Cancer Cooperative Group. The clinical database and the treatment guidelines of the Danish Breast Cancer Cooperative Group (DBCG); its 30-years experience and future promise. Acta Oncol. 2008;47(4):506-24. doi: 10.1080/02841860802059259. PMID 18465317
- [Background] Knoop AS, Knudsen H, Balslev E, Rasmussen BB, Overgaard J, Nielsen KV, Schonau A, Gunnarsdottir K, Olsen KE, Mouridsen H, Ejlertsen B; Danish Breast Cancer Cooperative Group. retrospective analysis of topoisomerase IIa amplifications and deletions as predictive markers in primary breast cancer patients randomly assigned to cyclophosphamide, methotrexate, and fluorouracil or cyclophosphamide, epirubicin, and fluorouracil: Danish Breast Cancer Cooperative Group. J Clin Oncol. 2005 Oct 20;23(30):7483-90. doi: 10.1200/JCO.2005.11.007. PMID 16234514
- [Background] Ejlertsen B, Tuxen MK, Jakobsen EH, Jensen MB, Knoop AS, Hojris I, Ewertz M, Balslev E, Dano H, Vestlev PM, Kenholm J, Nielsen DL, Bechmann T, Andersson M, Cold S, Nielsen HM, Maae E, Carlsen D, Mouridsen HT. Adjuvant Cyclophosphamide and Docetaxel With or Without Epirubicin for Early TOP2A-Normal Breast Cancer: DBCG 07-READ, an Open-Label, Phase III, Randomized Trial. J Clin Oncol. 2017 Aug 10;35(23):2639-2646. doi: 10.1200/JCO.2017.72.3494. Epub 2017 Jun 29. PMID 28661759
- [Derived] Jensen MB, Balslev E, Knoop AS, Tuxen MK, Hojris I, Jakobsen EH, Cold S, Dano H, Glavicic V, Kenholm J, Ejlertsen B. Adjuvant Docetaxel and Cyclophosphamide With or Without Epirubicin for Early Breast Cancer: Final Analysis of the Randomized DBCG 07-READ Trial. J Clin Oncol. 2025 Feb;43(4):373-380. doi: 10.1200/JCO.24.00836. Epub 2024 Oct 23. PMID 39442040
- [Derived] Fei F, Messina C, Slaets L, Chakiba C, Cameron D, Bogaerts J, Bonnefoi H. Tumour size is the only predictive factor of distant recurrence after pathological complete response to neoadjuvant chemotherapy in patients with large operable or locally advanced breast cancers: a sub-study of EORTC 10994/BIG 1-00 phase III trial. Eur J Cancer. 2015 Feb;51(3):301-9. doi: 10.1016/j.ejca.2014.11.023. Epub 2015 Jan 8. PMID 25578377
- [Derived] Eckhoff L, Knoop A, Jensen MB, Ewertz M. Persistence of docetaxel-induced neuropathy and impact on quality of life among breast cancer survivors. Eur J Cancer. 2015 Feb;51(3):292-300. doi: 10.1016/j.ejca.2014.11.024. Epub 2014 Dec 22. PMID 25541155
- See also: Danish Breast Cancer Cooperative Group — http://www.dbcg.dk